CLINICAL TRIAL: NCT05981742
Title: Effects of Combined Metformin and Cabergoline in Comparison With Metformin Only Therapy on Ovarian and Hormonal Activities in Iraqi Patients With PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Responsible Party: Principal Investigator, Hayder Adnan Fawzi, Associate Professor, Al-Rasheed University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR2023101
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrom; hormones; endometrial resistive index; metformin; Cabergoline
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (M) (Active Comparator): 25 Patients administered Metformin (Glucophage) Tablets of 500 mg per oral twice daily for 90 days duration.
  Interventions: Drug: Metformin Hydrochloride 500 MG
- Group 2 (D) (Active Comparator): 25 Patients administered Cabergoline (Pergoline) Tablets of 0.5 mg dose per oral once weekly for 90 days duration.
  Interventions: Drug: Cabergoline 0.5 MG
- Group 3 (MD) (Active Comparator): 25 Patients administered Metformin (Glucophage) Tablets of 500 mg per oral twice daily and Cabergoline (Pergoline) Tablets of 0.5 mg dose per oral once weekly for 90 days duration.
  Interventions: Drug: Metformin Hydrochloride 500 MG + Cabergoline 0.5 MG

INTERVENTIONS:
Drug: Metformin Hydrochloride 500 MG — Brand name: (Glucophage) Tablets per oral / Twice daily / 90 days duration
  Arms: Group 1 (M)
Drug: Cabergoline 0.5 MG — Brand name: (Pergoline) Tablets per oral / single dose per week / 90 days duration
  Arms: Group 2 (D)
Drug: Metformin Hydrochloride 500 MG + Cabergoline 0.5 MG — Metformin Brand name: (Glucophage) Tablets per oral / Twice daily / 90 days duration
  Cabergoline Brand name: (Pergoline) Tablets per oral / single dose per week / 90 days duration
  Arms: Group 3 (MD)

SUMMARY:
The goal of this interventional Randomized clinical is to compare the effect of Metformin alone, Cabergoline alone and Metformin and Cabergoline in combination in a sample of Iraqi female patients with polycystic ovary syndrome. The main questions to answer are:

1. What are the effects of the tested regimens on Body mass index (BMI)?
2. What are the effects of the tested regimens on hormonal status?
3. What are the effects of the tested regimens on uterine artery resistive index ?
4. What are the effects of the tested regimens on some inflammatory markers?

Participants will be separated into two groups:

1. Group 1 (M): 25 Patients, Received Metformin 500mg per oral twice daily for 90 days duration.
2. Group 2 (D): 25 Patients, Received Dostinex (Pergolin) 0.5 mg per oral (single dose per/week).
3. Group 3 (MD): 25 Pateins, Received metformin 500 mg per oral twice daily for 90 days duration and Dostinex (Pergolin) as 0.5 mg per oral (single dose per/week).

Researchers will compare Group 1 (M), Group 2 (D), Group 3 (MD) to observe the effect of the tested treatment regimens on Body Mass Index, Hormonal status, uterine artery resistive index, and some inflammatory markers that are IL-18, Anti-GAD Antibody and GnRH Antibody.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years
* Diagnosed with Polycystic Ovarian Syndrome based on Rotterdam criteria
* Body Mass Index (BMI) < 40 Kg/m²

Exclusion Criteria:

* Age less than 18 years or more than 40 years
* Co-morbid conditions including (diabetes mellitus, essential hypertension, and thyroid disease)
* Patients planning for conception.
* Body Mass Index > 40 Kg/m²

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | at Baseline, and after 90 days
  Measured in Kg/m² as a part of hormone status changes analysis
Serum Anti-Müllerian hormone (AMH) | at Baseline, and after 90 days
  Measured in ng/mL as a part of hormone status changes analysis
Serum Testosterone | at Baseline, and after 90 days
  Measured in ng/mL as a part of hormone status changes analysis
Serum Luteinizing hormone (LH) | at Baseline, and after 90 days
  Measured in mIU/mL as a part of hormone status changes analysis
Serum Follicular Stimulating Hormone (FSH) | at Baseline, and after 90 days
  Measured in mIU/mL as a part of hormone status changes analysis
Serum Prolactin (PRL) | at Baseline, and after 90 days
  Measured in ng/mL as a part of hormone status changes analysis
Mean number of dominant follicles (DF) | at Baseline, and after 90 days
  Calculated by ultrasonography as a part of the ultrasonic analysis
Mean Resistive Index (RI) | at Baseline, and after 90 days
  Calculated by ultrasonography as a part of the ultrasonic analysis
Serum Anti-GAD antibody | at Baseline, and after 90 days
  Measured in ng/mL as a part of inflammatory markers analysis
Serum Anti-GnRH antibody | at Baseline, and after 90 days
  Measured in pg/mL as a part of inflammatory markers analysis
Serum IL-18 Level | at Baseline, and after 90 days
  Measured in pg/mL as a part of inflammatory markers analysis

CONTACTS AND LOCATIONS:
Overall Officials: Inas Naser Hamad, B.Sc. Pharmacy, Principal Investigator — University of Al-Qadisiyah; Sinaa Abdul Amir Kadhim, Ph.D Pharmacology, Study Director — University of Al-Qadisiyah; Hayder Adnan Fawzi, Ph.D Clinical Pharmacy, Study Chair — Al-Mustafa University College
Locations (1):
- Maternity and Pediatric Teaching Hospital, Al Qādisīyah, Al-Qādisiyyah Governorate, Iraq